CLINICAL TRIAL: NCT04300855
Title: Phase II Clinical Trial of Green Tea Catechins in Men on Active Surveillance (AS)
Brief Title: Clinical Trial of Green Tea Catechins in Men on Active Surveillance
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: MCC-20056; 1R01CA235032-01A1 (NIH)
Record Dates: First submitted 2020-03-05; First posted 2020-03-09 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer; Prostate Adenocarcinoma
Keywords: Prostate; Green Tea; Green Tea Catechins
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Sunphenon

STUDY DESIGN:
Intervention Model Description: Participants participating in the study will be randomized 2:1 (2 study agent: 1 placebo) to receive Sunphenon® 90D (405 mg EGCG BID) or placebo.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sunphenon® 90D (Experimental): Participants will be administered a standardized formulation of whole Green Tea Catechin for 24 months. The daily dose of Green Tea Catechin will be taken in divided doses, three capsules in the morning and 3 capsules in the evening, with food (within one hour of eating a substantial meal). On the day of monthly follow-up visit, capsules should be taken within 4 hours of visit and blood draw for required lab work. If the participant is scheduled to come in the afternoon, dose should be taken with lunch that day instead of with dinner for that day.
  Interventions: Drug: Sunphenon
- Placebo (Placebo Comparator): Participants will be administered a placebo for 24 months. The daily dose of placebo will be taken in divided doses, three capsules in the morning and 3 capsules in the evening, with food (within one hour of eating a substantial meal). On the day of monthly follow-up visit, capsules should be taken within 4 hours of visit and blood draw for required lab work. If the participant is scheduled to come in the afternoon, dose should be taken with lunch that day instead of with dinner for that day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sunphenon — The study agent will be administered in divided doses with food, three capsules twice a day (405 mg) for 24 months
  Other Names: Green Tea Catechin
  Arms: Sunphenon® 90D
Drug: Placebo — Matching placebo
  Arms: Placebo

SUMMARY:
This randomized double-blinded Phase II clinical trial will evaluate the bioavailability, safety, effectiveness and validate the mechanism by which a standardized formulation of whole Green Tea Catechin, (Sunphenon® 90D) containing 405 mgs vs. Placebo, administered for 24 months in a cohort of men with low to intermediate grade prostate managed on active surveillance

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Biopsy-proven (consisting of ≥ 12 tissue cores) adenocarcinoma of the prostate with cancer present in at least one biopsy core (TRUS or/and mpMRI/TRUS fusion), Gleason score (3+3) or predominant Gleason pattern 3 (3+4), ≤ 33% of biopsy cores, and ≤50% involvement of any biopsy core (Participant meets all criteria for Active Surveillance as determined by MD)
* Willing to start or continue on active surveillance
* Baseline/screening serum PSA <10 ng/mL
* No other prior treatment for PCa, including focal therapy
* ECOG performance status 0-1
* No history of renal or hepatic disease, including history of hepatitis B and C
* Meet hematological eligibility parameters (Neutrophil count ≥ 1,200/mm3 (≥1.2 k/μL), Stable platelet count ≥ 75,000/mm3 (≥ 75k/μL) Hepatic and renal function eligibility parameters, serum total Bilirubin ≤ULN (ULN: 1.2 mg/dl) (or ≤3.0 mg/dL for patients with Gilbert's syndrome), AST or ALT <1.5x ULN and Serum creatinine ≤1.5 x ULN
* Willing to abstain from consumption of any supplements containing GTC
* Willing to restrict tea consumption to less than three (3) servings of hot tea or three (3) servings of iced tea per week
* Willing to discontinue current vitamin/mineral supplement use and use one provided by study
* Willing to take study agent or placebo at the dose specified with meals.

Exclusion Criteria:

* Have had prior treatment for PCa by surgery, irradiation, local ablative (i.e., cryosurgery or high-intensity focused ultrasound), or androgen-deprivation therapy)
* Men who are currently treated or those treated in the past 3 months prior to day of randomization with 5- alpha-reductase inhibitors (e.g., finasteride, dutasteride)
* Participants who have PCa with distant metastases
* Participants who have been treated with: hormone therapy, immunotherapy, chemotherapy and/or radiation, for any malignancies within the past 2 years prior to registration.Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial. All patients with metastatic disease will be excluded
* Participants may not be receiving any other investigational agents
* History of allergic reactions attributed to tea or compounds of similar chemical or biologic composition to green tea extracts.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 115 (Actual)
Dates: Start 2020-08-21 (Actual); Primary Completion 2027-02-27 (Estimated); Study Completion 2027-02-27 (Estimated)

PRIMARY OUTCOMES:
Rate of Progression to Prostate Cancer (PCa) | 24 months
  Number of participants with clinical progression defined as a composite outcome on repeat prostate biopsy >33% of biopsy cores positive for cancer or >50% of any biopsy tissue core positive for cancer or adverse reclassification of Gleason sum >3+3 or >3+4 respectively at end of study biopsy

SECONDARY OUTCOMES:
Occurrence of Adverse Events per Study Arm | Base line to 24 months
  Safety of Green Tea Catechins (GTC) at daily dose (vs. Placebo) as indicated by incidence of adverse events and toxicities, monitored using Common Toxicity Criteria version 5.0, complete blood count (CBC), and complete metabolic panel (CMP) from baseline, month 6, month 12 and month 24 at end of trial, Liver toxicities (LFTs) from baseline, month 3, 6 and every 3 months until end of intervention
Adherence of Green Tea Catechins vs.Placebo | Baseline to 24 months
  Adherence based on pill counts and agent logs
Acceptability of Green Tea Catechins vs.Placebo | Baseline to 24 months
  Acceptability based on pill counts and agent logs
Change in (prostate-specific antigen) PSA and PSA kinetics | Baseline to 24 months
  PSA or PSA density and PSA doubling time at month 12 and at 24 months) from serum at baseline, 6, 12, 18 and month 24
Change in gene expression panel | Baseline to 24 months
  Asses change in gene expression panel (Decipher) and a set of 13 biomarker genes known to be overexpressed in PCa from baseline to end of study (EOS) using biopsy tissue
Proportion of men with no cancer | Baseline to 24 months
  Assess the proportion of men with no cancer in the post-intervention biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Nagi Kumar, PhD RD FADA, Principal Investigator — Moffitt Cancer Center
Locations (2):
- United States (2):
  - Moffitt Cancer Center, Tampa, Florida
  - University of Kansas Cancer Center, Westwood, Kansas

IPD SHARING:
Plan to Share IPD: Undecided